CLINICAL TRIAL: NCT02152839
Title: The Implementation of Novel 'Heavy' Water Techniques for Determining Modulation of Muscle Protein, DNA and Lipid Synthesis Due to Ageing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Physiological Society (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Physoc_D20
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
MeSH Terms: interventions — Resistance Training

ARMS (2):
- Old Unilateral Exercise (Experimental): Old individuals (65-75y) studied before and after 6 weeks of unilateral resistance exercise training
  Interventions: Behavioral: Resistance Exercise
- Young Unilateral Exercise (Experimental): Young Individuals (18-30y) studied before and after 6 weeks unilateral resistance exercise training
  Interventions: Behavioral: Resistance Exercise

INTERVENTIONS:
Behavioral: Resistance Exercise — 6 Weeks progressive unilateral resistance exercise, 3 times per week, 70% 1-RM, 6 x 8 Repetitions. 2 minutes rest between sets

SUMMARY:
Maintenance of body's skeletal muscle is key to a healthy older age. However, as we age we lose on average 1-2% of our muscle each year. In order to slow this loss we need to understand fully the mechanisms regulating muscle mass with ageing. In this project we aim to determine these mechanisms using a new novel technique of 'heavy' water ingestion, which will allow us to measure multiple aspects of skeletal muscle mass control during normal everyday activities in young and old individuals over a period of 6 weeks. We will also determine the influence of resistance exercise training during this period in offsetting declines in muscle with ageing using this method

ELIGIBILITY:
Inclusion Criteria:

* Young (18-30y) and old men (65-75y) who are generally healthy and recreationally active

Exclusion Criteria:

* Active cardiovascular disease
* Cerebrovascular disease including previous stroke, aneurysm (large vessel or intracranial)
* Respiratory disease including pulmonary hypertension or COPD
* Hyper/ hypo parathyroidism, hyper/ hypothyroidism, Cushing's disease, diabetes
* Active inflammatory bowel disease
* Renal disease
* Malignancy
* Recent steroid treatment (within 6 mo), or hormone replacement therapy
* Clotting dysfunction
* Musculoskeletal or neurological disorders
* Any disease requiring long-term drug prescriptions, including statins

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | 0-6 Weeks
  Comparison of muscle protein synthesis between young and older individuals and in response to 6 weeks unilateral exercise training

SECONDARY OUTCOMES:
Muscle Sub fractions | 0-6 week
  Comparison of different sub fractions involved in muscle mass regulation between young and older individuals and in response unilateral exercise training

OTHER OUTCOMES:
Muscle Functions | 0-6 Weeks
  Muscle Strength and power un young and older individuals in response to unilateral exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Philip Atherton, PhD, AFHEA, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital Medical School, Derby, United Kingdom

REFERENCES:
- [Derived] Brook MS, Wilkinson DJ, Tarum J, Mitchell KW, Lund JL, Phillips BE, Szewczyk NJ, Kadi F, Greenhaff PL, Smith K, Atherton PJ. Neither myonuclear accretion nor a myonuclear domain size ceiling is a feature of the attenuated hypertrophic potential of aged human skeletal muscle. Geroscience. 2023 Feb;45(1):451-462. doi: 10.1007/s11357-022-00651-y. Epub 2022 Sep 9. PMID 36083436